CLINICAL TRIAL: NCT06750965
Title: Epidemiological Characteristics Associated With Precursor Lesions of Multiple Myeloma Using Serum M Protein Screening: a Multi-center, Prospective Cohort Study.
Brief Title: Multi-center Screening for Serum M Protein
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Zhujiang multi-center
Record Dates: First submitted 2024-01-04; First posted 2024-12-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Monoclonal Gammopathy; Multiple Myeloma; M-protein
Keywords: M-protein
MeSH Terms: conditions — Paraproteinemias; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Physical examination population （Screening stage）: Subjects of different age groups in different sub-centers nationwide for physical examination
  Interventions: Diagnostic Test: Serum M protein screening
- Positive subjects for M-protein screening （Follow up stage）: Each sub-center will include subjects who are positive for M protein screening based on their actual situation.
  Interventions: Diagnostic Test: Serum M protein screening
- Negative control subjects （Follow up stage）: Each sub-center matched control subjects with negative M protein detection by age and gender parameter 1:1.
  Interventions: Diagnostic Test: Serum M protein screening

INTERVENTIONS:
Diagnostic Test: Serum M protein screening — Using highly sensitivity test to screen serum M protein of all participants.

SUMMARY:
This study aims to utilize a highly sensitive method for detecting M protein in serum to examine the prevalence of M protein in various age groups of individuals aged over 30 who underwent physical examinations in different regions of China. Furthermore, the study seeks to analyze the relationship between physical examination indicators and the presence of serum M protein (as measured by relative intensity) in the study participants at the time of enrollment. Additionally, a 5-year follow-up period will be employed to observe the association between annual physical examination indicators and clinical outcomes in subjects identified with positive/negative serum M protein screening.

DETAILED DESCRIPTION:
Monoclonal gammopathy (MG) is an asymptomatic premalignant clonal proliferation of plasma cells. The onset of this condition is typically concealed and often serendipitously discovered by patients through various clinical symptoms or the detection of monoclonal gamma globulin (M protein) using protein electrophoresis during disease evaluation. Although monoclonal gammopathy of unknown significance (MGUS) usually remains asymptomatic, it can progress to multiple myeloma (MM) over time. With the aging population, the prevalence of MGUS continues to rise among the general population. Therefore, it is crucial to screen individuals over the age of 50, or even younger, for serum M protein.

Currently, the investigators have established a highly sensitive and high-throughput flight mass spectrometry-based method for detecting M protein. In this study, the investigators aim to conduct a nationwide, multicenter, and prospective follow-up study involving participants from the general physical examination population. The study's objective is to investigate the epidemiological characteristics of targeted serum M protein screening for precancerous lesions in multiple myeloma. The investigators will assess the proportion of individuals with positive serum M protein in different age groups within the physical examination population aged over 30 from various regions in China. Additionally, the investigators will analyze the correlation between physical examination indicators such as liver and kidney function and the presence of serum M protein. Furthermore, the investigators will analyze the relationship between serum M protein levels, disease progression, and other clinical outcomes through annual follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

(1) Screening stage

1. Over 30 years old.
2. Volunteer to participate in this study and sign an informed consent form.

(2) Follow up stage

1. According to previous studies, a positive rate of 5% -8% was found in subjects with positive M protein screening. Each sub center included approximately 50-80 positive subjects based on actual conditions. At the same time, control subjects with negative M protein testing were matched by age and gender parameter 1:1.
2. Volunteer to participate in the follow-up phase of the study and sign an informed consent form.

Exclusion Criteria:

(1) Screening stage

1) Previously diagnosed with hematological diseases such as plasma cell or other B lymphocyte proliferative diseases.

Culling criteria:

1. Samples with incomplete or untraceable subject data.
2. Unqualified samples: including serum samples with severe hemolysis, fatty blood or jaundice, insufficient sample, and samples not stored as required.
3. The subject requested to withdraw from the study midway.
4. Duplicate samples of subjects at the same time point.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population is a physical examination population aged over 30 and of different age groups from different regions of China. This study selected the study population as the research object based on inclusion, exclusion, and culling criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive rate of serum M protein | 1 year
  In the stage of enrollment of this cross-sectional study, investigate the positive rate of serum M protein in subjects of different age groups in different sub-centers across the country, and analyze the correlation between M protein positive and physical examination indicators.

SECONDARY OUTCOMES:
The correlation between serum M protein positivity and related symptoms and indicators | Five years
  At every follow-up time points, to observe the correlation between serum M protein positivity and related symptoms and indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Zhou, Professor, Study Chair — Zhujiang Hospital

IPD SHARING:
Plan to Share IPD: No